CLINICAL TRIAL: NCT02142244
Title: Infrared Fluorescence Guided Surgery for Sentinel Node Identification in Cutaneous Melanoma
Brief Title: Fluorescence Surgery for Sentinel Node Identification in Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BCHNIR01
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-09

CONDITIONS: Melanoma; Lymph Node Metastasis
Keywords: Sentinel node biopsy; Near infra red light; Indocyanine green; micrometastasis
MeSH Terms: conditions — Melanoma; Lymphatic Metastasis; Neoplasm Micrometastasis | interventions — Sentinel Lymph Node Biopsy; Fluorescence; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Near infra red sentinel node biopsy (Experimental): Sentinel node biopsy adding indocyanine green injection at the tumor/biopsy site during the surgical procedure to the standard technique (blue die and lymph scintigraphy) and near infra red light for fluorescence. The indocyanine green saline solution - 5mg diluted in 10ml. will be injected in 4 points around the biopsy site - 4ml each - total 0.8mg - single procedure.Near infra red lens and camera will be used to detect the fluorescence and localize the sentinel node for biopsy.
  Interventions: Procedure: Near infra red sentinel node biopsy; Drug: Indocyanine green; Device: Intraoperative Near-Infrared Imaging System

INTERVENTIONS:
Procedure: Near infra red sentinel node biopsy — Explicated in the protocol arm
  Other Names: Sentinel node biopsy with fluorescence
Drug: Indocyanine green — Explicated in the protocol arm
Device: Intraoperative Near-Infrared Imaging System — Explicated in the protocol arm
  Other Names: Photodynamic Eye (PDE); Pulsion; MiniFlare; The Flare Foundation

SUMMARY:
Sentinel node biopsy is a surgical procedure used to find melanoma lymph node metastasis (i.e. groin/axilla) in very early stages. This study aims to add a new technology over the standard procedure - a fluorescent contrast (indocyanine green) using special light (near infra-red) - looking for more precise diagnosis of the presence of the lymph node metastasis.

DETAILED DESCRIPTION:
The main objectives of this study is perform a new technique added to the usual procedure for sentinel lymph node biopsy for cutaneous melanoma. The fluorescence surgery consists in a injection of indocyanine green around the primary tumor, or, when already excised (excisional biopsy), the biopsy site at the beginning of the surgery. Patient performs, in a standard fashion, the lymph scintigraphy prior the surgery and is injected at the same time a blue die similarly the indocyanine green. Immediately after the indocyanine infusion, the injection site is massaged and a near infra red light (NIR) is focused over it. An appropriated infra red camera is positioned over the lymphatic pathway, searching for the fluorescence and localizing the sentinel node at the basin. The skin is opened and the sentinel node is resected. The success or not in localizing the sentinel node is pointed and the standard techniques are applied - gamma probe and surgical location of a blue lymph node. All sentinel node characteristics are noted as number, which technic identified it, time, location. Later information will be gathered as histological status, surgical complications, recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for sentinel node biopsy in standard care

Exclusion Criteria:

* Previous neoplasia
* Previous surgery or scar in the lymph node basin or primary tumor, except primary tumor biopsy
* Local recurrence
* Hypersensibility or allergy history to indocyanine or Iodine-based contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Sensibility of the sentinel node biopsy | Time of surgery
  The successful rate of the sentinel node localization and biopsy. The standard technique and the experimental one will be assessed

SECONDARY OUTCOMES:
Specificity of the sentinel node biopsy | 60 months
  The false negative sentinel node biopsy rate. The proportion of patients submitted to the procedure with histological negative biopsy, presenting lymph node metastasis at follow up.

OTHER OUTCOMES:
Overall survival | 60 months
Disease free survival | 60 months
  Presence and time to disease recurrence or not
Specific cancer survival | 60 months
  Specific melanoma survival

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius L Vazquez, Ph.D., Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

REFERENCES:
- [Background] Tanaka E, Choi HS, Fujii H, Bawendi MG, Frangioni JV. Image-guided oncologic surgery using invisible light: completed pre-clinical development for sentinel lymph node mapping. Ann Surg Oncol. 2006 Dec;13(12):1671-81. doi: 10.1245/s10434-006-9194-6. Epub 2006 Sep 29. PMID 17009138
- [Background] Frangioni JV. New technologies for human cancer imaging. J Clin Oncol. 2008 Aug 20;26(24):4012-21. doi: 10.1200/JCO.2007.14.3065. PMID 18711192
- [Background] Namikawa K, Yamazaki N. Sentinel lymph node biopsy guided by indocyanine green fluorescence for cutaneous melanoma. Eur J Dermatol. 2011 Mar-Apr;21(2):184-90. doi: 10.1684/ejd.2010.1237. PMID 21498148
- [Background] van der Vorst JR, Schaafsma BE, Verbeek FP, Swijnenburg RJ, Hutteman M, Liefers GJ, van de Velde CJ, Frangioni JV, Vahrmeijer AL. Dose optimization for near-infrared fluorescence sentinel lymph node mapping in patients with melanoma. Br J Dermatol. 2013 Jan;168(1):93-8. doi: 10.1111/bjd.12059. PMID 23078649